CLINICAL TRIAL: NCT03767504
Title: An Open Label Study to Evaluate the Effect and Tolerance of Musclin™ (Thymol) in Healthy Subjects
Brief Title: A Study to Evaluate the Effect and Tolerance of Musclin™ (Thymol) in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INNV-MS1000-001
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Thymol

STUDY DESIGN:
Intervention Model Description: Open label, single arm, ascending dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musclin (Experimental): Thymol based dietary supplement
  Interventions: Dietary Supplement: Thymol

INTERVENTIONS:
Dietary Supplement: Thymol — Musclin - a dietary supplement: 2 capsules (20 mg thymol per capsule) BID with a meal for 30 days increased to 4 capsules for an additional 30 days.
  Other Names: Musclin

SUMMARY:
This study is to evaluate the effect and tolerance of a thymol containing dietary supplement, Musclin, in healthy adults.

DETAILED DESCRIPTION:
This study will be an open label, uncontrolled, ascending dose clinical trial to assess the tolerance and effect of orally ingested Musclin, 20 mg thymol per capsule, in healthy adult subjects. In addition, this study will evaluate whether Musclin has an effect on creatine kinase and myostatin levels. The study will aim to enroll 20 consenting men and women. Consented subjects will ingest 2 capsules of Musclin daily for 30 days and increase to 4 capsules daily for an additional 30 days . Physical assessments and biological samples will be collected at baseline (day 0) and at end of treatment (d 60). Surveys to include reported stamina and energy levels will be collected at baseline, prior to increased dosage (d 30) and end of treatment period. Risk to participants is expected to be minimal and will be outlined through an informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer > 40 years (adult)
2. Systolic blood pressure 90-140 mmHg upon screening
3. Subject has provided written informed consent
4. Subject is willing to undergo the procedures outlined in this study
5. Subjects BMI is within 18-28.
6. Subjects of childbearing potential must use a hormonal method of birth control, single-barrier method or a double-barrier method of birth control throughout the study or be documented as medically sterile.

Exclusion Criteria:

1. Subject has clinically significant deviation from normal in any organ system.
2. Subject has a clinically significant deviation from normal in any laboratory test except high cholesterol.
3. Pregnant, breastfeeding, or planned pregnancy during the study duration.
4. Known liver, renal or muscle diseases.
5. History of hypertensive or currently taking anti-hypertensive medications.
6. Presence or history of specific heart conditions.
7. Currently taking anti-thyroid or thyroid replacement medications.
8. Currently taking any creatinine kinase lowering drug or supplement.
9. Use of investigational drug within the previous 30 days.
10. Use of herbal supplements, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within 2 weeks prior to initial dosing.
11. Known allergies or intolerance to ingredients in Musclin™
12. Any condition which would interfere with the subject's ability to provide informed consent, to comply with study instructions, or which might confound the interpretation of the study results.

    -

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-02-13 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse events as a measure of tolerance | Day 60 (End of Study)
Change in creatinine kinase | Day 1(Baseline) to Day 60 (End of Study)
  Change in creatinine kinase measured in U/L
Change in myostatin levels | Day 1(Baseline) to Day 60 (End of Study)
  Change in myostatin will be measured by blood samples using ELISA method.

SECONDARY OUTCOMES:
Changes in weight | Day 1(Baseline) to Day 60 (End of Study)
  Effect of supplement on weight (lbs)
Change in cholesterol levels | Day 1(Baseline) to Day 60 (End of Study)
  Effect of supplement on cholesterol levels
Number, type, and severity of adverse events | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Palm Beach Research Center, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No